CLINICAL TRIAL: NCT02078648
Title: A Phase 1/2 Study of SL-701, a Subcutaneously Injected Multivalent Glioma-Associated Antigen Vaccine, in Adult Subjects With Recurrent Glioblastoma Multiforme
Brief Title: Safety and Efficacy Study of SL-701, a Glioma-Associated Antigen Vaccine To Treat Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STML-701-0114
Record Dates: First submitted 2014-02-20; First posted 2014-03-05 (Estimated); Results first posted 2023-12-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Adult Brain Glioblastoma; Glioblastoma Multiforme
Keywords: Glioma Associated Antigen; Vaccine; Adult; Recurrent Glioblastoma; Immunotherapy
MeSH Terms: conditions — Glioblastoma | interventions — poly ICLC; Polylysine; Carboxymethylcellulose Sodium; Bevacizumab; Granulocyte-Macrophage Colony-Stimulating Factor; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SL-701 + GM-CSF + Imiquimod (Experimental): Participants will receive SL-701 with the vaccine adjuvants granulocyte macrophage-colony stimulating factor (GM-CSF) injection and imiquimod topical cream.
  A complete dose of study drug consists of the administration of a sequence of 3 agents, SL-701 emulsion SC injection, GM-CSF SC injection, and imiquimod topical cream, within a 5-minute time frame. Topical application of imiquimod cream at the injection site is repeated at 24 hours after each SL-701 emulsion injection. For each participant, SL-701 emulsion (SL-701 in Montanide) will be administered by SC injection beginning on Day 1 with imiquimod topical cream 5% applied immediately (within 5 minutes of SL-701 emulsion injection) to the SL-701 emulsion injection site.
  In addition to the SL-701 emulsion injection, the participant will receive a SC injection of GM-CSF 150 μg close to the injection site of SL-701 emulsion. An additional dose of imiquimod cream will be applied at the same site by the participant 24 hours later.
  Interventions: Drug: SL-701 + GM-CSF; Drug: Imiquimod
- SL-701; poly-ICLC 1.6 mg; bevacizumab (Experimental): SL-701 emulsion and the adjuvant poly-ICLC will be administered twice weekly for the initial 2 weeks, every 7 days during the subsequent 3 doses, and subsequently every 14 days for the subsequent 9 doses (16 doses total) through Week 22, and every 4 weeks thereafter. Bevacizumab will be administered every 2 weeks, subsequent to the administration of SL-701/poly-ICLC.
  Interventions: Drug: SL-701; poly-ICLC (polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethyl cellulose); Drug: Bevacizumab

INTERVENTIONS:
Drug: SL-701; poly-ICLC (polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethyl cellulose) — 1.0 mL injection taken from 0.7 mL of SL-701 mixed at a 1:1 (v/v) ratio with 0.7 mL of Montanide. Preferred site of SC injection is in the right or left upper arms.
  Within 20 minutes following the administration of the SL-701 emulsion, poly-ICLC should be administered as an IM injection in the same extremity (within 3 cm whenever possible) as was administered the SL-701 (deltoid muscle, unless contraindicated).
  Other Names: Avastin
  Arms: SL-701; poly-ICLC 1.6 mg; bevacizumab
Drug: Bevacizumab — Following the administration of SL-701 and poly-ICLC, bevacizumab will be administered IV at a dose of 10 mg/kg. Bevacizumab infusions may occur over 30, 60 or 90 minutes in accordance with institutional practices and guidelines.
  Arms: SL-701; poly-ICLC 1.6 mg; bevacizumab
Drug: SL-701 + GM-CSF — 1.0 mL injection taken from 0.7 mL of SL-701 mixed at a 1:1 (v/v) ratio with 0.7 mL of Montanide. Preferred site of SC injection is in the right or left upper arms.
  150 μg GM-CSF should be administered as a SC injection immediately after SL-701 emulsion administration and within 1 cm from the center of the SL-701 emulsion injection site.
  Arms: SL-701 + GM-CSF + Imiquimod
Drug: Imiquimod — Within 5 minutes following the administration of the SL-701 emulsion, approximately 125 mg of imiquimod cream will be applied topically on the injection site. The imiquimod cream should be rubbed in until the cream is no longer visible.
  Arms: SL-701 + GM-CSF + Imiquimod

SUMMARY:
The purpose of this study is to determine the safety and efficacy of SL-701 as a treatment for recurrent glioblastoma multiform (GBM).

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 1/2 study evaluating the efficacy and safety of SL-701 as a treatment for recurrent GBM, divided into 2 stages. Seventy-four (74) participants were treated in the study, 46 in Stage 1 and 28 in Stage 2, men and women at least 18 years of age, all of whom showed unequivocal evidence of either a first tumor recurrence or progression during or following an initial treatment regimen before enrollment in this study. At least 54 of the 74 treated participants had measurable disease based on contrast-enhanced magnetic resonance imaging or computed tomography scans.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Histologically confirmed GBM or World Health Organization (WHO) Grade IV variants (gliosarcoma, glioblastoma with oligodendroglial features, or giant cell glioblastoma).
* Unequivocal evidence of a first tumor recurrence or progression on the initial treatment regimen (prior to enrollment on this study), consisting of surgical intervention (biopsy and/or resection), radiation, and temozolomide chemotherapy, as assessed by MRI or CT scan of the brain with or without contrast within 14 days prior to the start of SL-701. If receiving corticosteroids, the dose must be stable or decreasing for at least 5 days prior to the scan. Participants unable to undergo MRI because of non-compatible devices can be enrolled, provided CT scans are obtained and are of sufficient quality. For each participant, the same imaging technique should be performed throughout the study, for purposes of assessing tumor response or PD.
* For participants who have undergone resection of recurrent or progressive tumor prior to study enrollment, the following conditions must apply:

  * Recovery from the effects of surgery.
  * Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, an MRI should be performed:

    * No later than 96 hours (h) in the immediate post-operative period; or
    * At least 4 weeks post-craniotomy (7 days for stereotactic biopsy), within 14 days prior to the start of SL-701, and on a corticosteroid dosage that has been stable or decreasing for at least 5 days.
* Participants who have not had resection of recurrent or progressive disease must have measurable disease.
* At least 56 of the approximately 76 participants treated must have measurable disease, defined as at least one, contrast-enhancing lesion measuring at least 1 cm in 2 planes (axial, coronal, or sagittal).
* No evidence of hemorrhage on the baseline MRI or CT scan other than those that are Grade ≤ 1 and either post-operative or stable on at least two consecutive scans.
* Recovery from prior therapy toxicity, defined as resolution of all treatment-related adverse events (AEs) to Grade ≤ 1 or pre-treatment baseline (except alopecia and lymphopenia).
* At least 12 weeks from prior radiotherapy to the start of SL-701 unless there is new enhancement outside of the radiation field or unequivocal histopathologic evidence of recurrent tumor subsequent to radiotherapy.
* No chemotherapy or investigational agent for at least 3 weeks prior to the start of SL-701.
* Human leukocyte antigen (HLA)-A2 positive.
* A tumor tissue sample is provided for immunohistochemical analysis of relevant antigens, immune markers and potential prognostic factors. Preferably a paraffin block or 10-12 unstained slides will be submitted prior to study entry. Participants for whom tumor samples are unavailable or inadequate are permitted to participate in the study; however, the absence of available/adequate tumor specimen must be documented.
* Karnofsky performance status (KPS) score ≥ 70%.
* Adequate organ function, including the following:

  * Absolute neutrophil count (ANC) ≥ 1,000/μL, platelets ≥ 100,000/μL.
  * Serum creatinine < 1.5 × the upper limit of normal (ULN).
  * Bilirubin < 1.5 × ULN.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 × ULN.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to the start of SL-701 treatment.
* Female participants of childbearing potential and sexually active male participants must agree to use an acceptable form of contraception for heterosexual activity (that is, oral contraceptives, double barrier methods, hormonal injectable, transdermal, or implanted contraceptives, tubal ligation, or vasectomy of their sexual partner(s) for > 40 days before Screening, during the study, and for 60 days after the last dose of study drug. Men should not donate semen during the study and for 60 days after the last dose of study drug.
* Female participants without childbearing potential (spontaneous amenorrhea for > 12 months or surgically sterilized by tubal ligation, hysterectomy, or bilateral oophorectomy > 6 months before Screening) are eligible for inclusion without contraceptive use restriction.
* Able and willing to comply with protocol requirements, in the opinion of the investigator.
* A written and voluntarily signed informed consent must be obtained from the participant or legally authorized representative, in accordance with local regulations, before the initiation of any study related procedures. The participant or legally authorized representative must be able to read and understand the informed consent form (ICF).

Exclusion Criteria:

* Prior cancer chemotherapy, bevacizumab (or other vascular endothelial growth factor [VEGF]/VEGF receptor [VEGFR]-directed agent), or an investigational agent for recurrent/progressive GBM or prior bevacizumab as part of initial therapy (prior chemotherapy or investigational agents are permitted as part of initial therapy; VEGF/VEGFR-directed agents are not permitted).
* Contrast-enhancing tumor that is any of the following:

  * Multi-focal (defined as two separate areas of contrast enhancement measuring at least 1 cm in 2 planes that are not contiguous on either fluid-attenuated inversion recovery (FLAIR) or T2 sequences);
  * Associated with either diffuse subependymal or leptomeningeal dissemination; or
  * ≥ 4 cm in any dimension.
* Requirement of systemic corticosteroid therapy > 4 mg/day of dexamethasone or equivalent or requirement of increasing dose of systemic corticosteroids during the 7 days prior to the start of SL-701 treatment.
* Surgical resection or major surgical procedure within 4 weeks prior to the start of SL-701, or stereotactic biopsy within 7 days prior to the start of SL-701.
* Radiation therapy, local therapy (except for surgical re-resection), or systemic therapy following first recurrence/progressive disease. Excluded local therapies include stereotactic radiation boost, implantation of carmustine biodegradable wafers (Gliadel), intratumoral or convection-enhanced delivery administered agents, etc.
* Active infection requiring intravenous antibiotics.
* History of cancer (other than GBM) within the past 2 years that has metastatic or local recurrence potential and could negatively impact survival and/or potentially confound tumor response assessments within this study.
* Clinically significant cardiovascular disease (for example, uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction or stroke within 6 months of study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication).
* Known immunosuppressive disease or active systemic autoimmune disease such as systemic lupus erythematosus, human immunodeficiency virus infection, Hepatitis B, or Hepatitis C, or has taken an immunosuppressive agent within 4 weeks prior to the start of SL-701 treatment. Participants with vitiligo, type 1 diabetes mellitus, hypothyroidism due to autoimmune condition only requiring hormone replacement therapy, psoriasis not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Any condition which in the investigator's opinion makes the participant unsuitable for study participation.
* Requires therapeutic anticoagulation with warfarin at baseline; participants must be off warfarin or warfarin-derivative anti-coagulants for at least 7 days prior to starting study drug; however, therapeutic or prophylactic therapy with low-molecular weight heparin is allowed.
* Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of start of study drug.
* Has evidence of intratumoral or peritumoral hemorrhage on baseline MRI scan other than those that are ≤Grade 1 and either post-operative or stable on at least 2 consecutive MRI scans
* Has gastrointestinal bleeding or any other hemorrhage/bleeding event National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) >Grade 3 within 6 months of start of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - George Washington University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Baylor Charles A Sammons Cancer Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- SL-701 + GM-CSF + Imiquimod: Participants received SL-701 with the vaccine adjuvants granulocyte-macrophage colony-stimulating factor (GM-CSF) injection and imiquimod topical cream.
  A complete dose of study drug consisted of the administration of a sequence of 3 agents, SL-701 emulsion subcutaneous (SC) injection, GM-CSF SC injection, and imiquimod topical cream, within a 5-minute time frame. Topical application of imiquimod cream at the injection site was repeated at 24 hours (h) after each SL-701 emulsion injection. For each participant, SL-701 emulsion (SL-701 in Montanide) was administered by SC injection beginning on Day 1 with imiquimod topical cream 5% applied immediately (within 5 minutes after SL-701 emulsion injection) to the SL-701 emulsion injection site.
  In addition to the SL-701 emulsion injection, the participant received a SC injection of GM-CSF 150 micrograms (μg) close to the injection site of SL-701 emulsion (immediately following the SL-701 emulsion injection, before the application of topical imiquimod). An additional dose of imiquimod cream was applied at the same site by the participant 24 h later.
- SL-701 + Poly-ICLC + Bevacizumab: SL-701 emulsion and the adjuvant polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethyl cellulose (poly-ICLC) were administered twice weekly for the initial 2 weeks, every 7 days during the subsequent 3 doses, and subsequently every 14 days for the subsequent 9 doses (16 doses total) through Week 22, and every 4 weeks thereafter. Bevacizumab was administered every 2 weeks, after the administration of SL-701/poly-ICLC.
  SL-701: Within 20 minutes following the administration of the SL-701 emulsion, poly-ICLC was administered as an intramuscular (IM) injection in the same extremity (within 3 centimeters [cm] whenever possible) as was administered the SL-701 (deltoid muscle, unless contraindicated).
  Bevacizumab: Following the administration of SL-701 and poly-ICLC, bevacizumab was administered intravenously (IV) at a dose of 10 milligrams/kilogram (mg/kg). Bevacizumab infusions occurred over 30, 60 or 90 minutes in accordance with institutional practices and guidelines.
Period: Overall Study
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Started | 46 | 28
Received At Least 1 Dose of Study Drug (Intent-to-Treat Population) | 46 | 28
Completed | 0 | 0
Not Completed | 46 | 28
Not completed — Unequivocal Evidence of Disease Progression | 36 | 13
Not completed — Adverse Event | 0 | 1
Not completed — General Deterioration in Performance Status Without Radiographic Evidence of Disease Progression | 1 | 4
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Investigator Decision | 5 | 7
Not completed — Death | 1 | 1
Not completed — Undefined | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Groups:
- SL-701 + GM-CSF + Imiquimod: Participants received SL-701 with the vaccine adjuvants GM-CSF injection and imiquimod topical cream.
  A complete dose of study drug consisted of the administration of a sequence of 3 agents, SL-701 emulsion SC injection, GM-CSF SC injection, and imiquimod topical cream, within a 5-minute time frame. Topical application of imiquimod cream at the injection site was repeated at 24 h after each SL-701 emulsion injection. For each participant, SL-701 emulsion (SL-701 in Montanide) was administered by SC injection beginning on Day 1 with imiquimod topical cream 5% applied immediately (within 5 minutes after SL-701 emulsion injection) to the SL-701 emulsion injection site.
  In addition to the SL-701 emulsion injection, the participant received a SC injection of GM-CSF 150 μg close to the injection site of SL-701 emulsion (immediately following the SL-701 emulsion injection, before the application of topical imiquimod). An additional dose of imiquimod cream was applied at the same site by the participant 24 h later.
- SL-701 + Poly-ICLC + Bevacizumab: SL-701 emulsion and the adjuvant poly-ICLC were administered twice weekly for the initial 2 weeks, every 7 days during the subsequent 3 doses, and subsequently every 14 days for the subsequent 9 doses (16 doses total) through Week 22, and every 4 weeks thereafter. Bevacizumab was administered every 2 weeks, after the administration of SL-701/poly-ICLC.
  SL-701: Within 20 minutes following the administration of the SL-701 emulsion, poly-ICLC was administered as an IM injection in the same extremity (within 3 cm whenever possible) as was administered the SL-701 (deltoid muscle, unless contraindicated).
  Bevacizumab: Following the administration of SL-701 and poly-ICLC, bevacizumab was administered IV at a dose of 10 mg/kg. Bevacizumab infusions occurred over 30, 60 or 90 minutes in accordance with institutional practices and guidelines.
- Total: Total of all reporting groups
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab | Total
Number analyzed (Participants) | 46 | 28 | 74
Age, Continuous [Mean (Full Range); unit: years] | 52.9 [23.9 to 71.6] | 60.0 [25.7 to 79.1] | 55.6 [23.9 to 79.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 30 | 18 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 39 | 25 | 64
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 40 | 25 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter squared] — Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701 and with the last non-missing assessment taken prior to administration of the first SL-701 injection.
  kilogram/meter squared
    number analyzed (Participants) | 41 | 24 | 65
    (all) | 28.3 (6.0) | 29.4 (6.2) | 28.7 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Regimen-limiting Toxicity (RLT)
Description: RLT included any events that occurred anytime through the first 12 doses of study treatment that were considered possibly, probably, or definitely related to investigational therapy and ranged from Grade ≥3 bronchospasm or Grade 2 bronchospasm that did not resolve within 24 hours despite appropriate medical treatment to cerebral edema associated with severe clinical manifestations (Grade 4) that were considered related to study therapy by the investigator.
Time Frame: Approximately 24 weeks
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Count of Participants; unit: Participants
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
Participants | 0 | 0

2. Primary Outcome: Number of Participants Experiencing Sudden or Unexpected Death Related to SL-701 or SL-701 in Combination With Bevacizumab
Description: A safety review occurred following each sudden or unexpected death that was not considered by the investigator to be a disease-related mortality and was considered to be related to SL-701.
Time Frame: Day 1 through Month 12
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Count of Participants; unit: Participants
Groups:
- SL-701 + GMCSF + Imiquimod: Participants received SL-701 with the vaccine adjuvants GM-CSF injection and imiquimod topical cream.
  A complete dose of study drug consisted of the administration of a sequence of 3 agents, SL-701 emulsion SC injection, GM-CSF SC injection, and imiquimod topical cream, within a 5-minute time frame. Topical application of imiquimod cream at the injection site was repeated at 24 h after each SL-701 emulsion injection. For each participant, SL-701 emulsion (SL-701 in Montanide) was administered by SC injection beginning on Day 1 with imiquimod topical cream 5% applied immediately (within 5 minutes after SL-701 emulsion injection) to the SL-701 emulsion injection site.
  In addition to the SL-701 emulsion injection, the participant received a SC injection of GM-CSF 150 μg close to the injection site of SL-701 emulsion (immediately following the SL-701 emulsion injection, before the application of topical imiquimod). An additional dose of imiquimod cream was applied at the same site by the participant 24 h later.
Arm/Group | SL-701 + GMCSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
Participants | 0 | 0

3. Primary Outcome: Overall Survival at 12 Months (OS-12)
Description: OS-12 was defined as the number of participants surviving at 12 months after the first injection of SL-701 and was calculated using the Clopper-Pearson Method.
Time Frame: Up to 12 months
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Count of Participants; unit: Participants
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
Participants | 20 | 14

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was the percentage of participants who had at least 1 overall tumor response of complete response (CR) or partial response (PR) documented on 2 consecutive magnetic resonance images (MRIs) ≥4 weeks apart by modified response assessment in neuro-oncology (RANO) criteria.
Time Frame: 3 years
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
percentage of participants | 2.2 [0.1 to 9.9] | 14.3 [5.0 to 29.8]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was the percentage of participants whose best response was either CR, PR, or stable disease (SD) documented on 2 consecutive MRIs ≥4 weeks apart by modified RANO criteria.
Time Frame: 3 years
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
percentage of participants | 21.7 [10.9 to 36.4] | 53.6 [33.9 to 72.5]

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the time from the date measurement criteria were first met for objective response (either CR or PR) until the first date that the criteria for progressive disease (PD) was met, or death due to any cause, whichever occurred first, by modified RANO. If a participant did not progress or die after a response of CR or PR, then the participant's DoR was censored at the date of the participant's last tumor assessment. Only participants who attained a confirmed response of either CR or PR were included in the estimation of DoR (calculated using the Kaplan-Meier method).
Time Frame: 3 years
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Median (90% Confidence Interval); unit: month
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 1 | 4
month | NA [NA to NA] — Values were non-estimable (insufficient number of participants with events). | 8.8 [NA to NA] — Values were non-estimable (high censoring rates).

7. Secondary Outcome: Duration of Disease Control (DDC)
Description: DDC was defined as the time from the date measurement criteria were first met for objective response (either CR, PR, or SD) until the first date that the criteria for PD were met, or death due to any cause, whichever occurs first, by modified RANO. If a participant did not progress or die after a response of CR, PR or SD, then the participant's DDC was censored at the date of the participant's last tumor assessment. Only participants who attained a confirmed response of either CR, PR or SD were included in the estimation of DDC.
Time Frame: 3 years
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 10 | 15
month | 9.2 [3.8 to NA] — Values were non-estimable (insufficient number of participants with events). | 8.8 [3.7 to NA] — Values were non-estimable (insufficient number of participants with events).

8. Secondary Outcome: Progression-free Survival at 6 Months (PFS-6)
Description: PFS-6 was defined as the time from the date of the first injection of SL-701 to the date of disease progression or death from any cause, whichever occurred first, by modified RANO. Participants who had not progressed or died at the time of the analysis were censored at the date of their latest tumor assessment or survival assessment.
Time Frame: Up to 6 months
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
month | 1.9 [1.8 to 2.7] | 5.6 [3.3 to NA] — Values were non-estimable (insufficient number of participants with events).

9. Secondary Outcome: Progression-free Survival at 12 Months (PFS-12)
Description: PFS-12 was defined as the time from the date of the first injection of SL-701 to the date of disease progression or death from any cause, whichever occurred first, by modified RANO. Participants who had not progressed or died at the time of the analysis were censored at the date of their latest tumor assessment.
Time Frame: Up to 12 months
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
month | 1.9 [1.8 to 2.7] | 5.6 [3.6 to 10.0]

10. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of the first injection of SL-701 to the date of disease progression or death from any cause, whichever occurred first, by modified RANO. Participants who had not progressed or died at the time of the analysis were censored at the date of their latest tumor assessment.
Time Frame: 3 years
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
month | 1.9 [1.8 to 2.7] | 5.6 [3.6 to 10.0]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was the time from the date of the first SL-701 injection to the date of death from any cause. If a participant did not die during the study, the participant's overall survival time was censored at the date at which the participant was last known to be alive.
Time Frame: 3 years
Population: Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
Number analyzed (Participants) | 46 | 28
month | 10.9 [8.2 to 12.0] | 11.7 [7.1 to NA] — Values were non-estimable (insufficient number of participants with events).

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: up to 3 years; Serious and Other Adverse Events: up to Month 12; Survival (PFS, OS), ORR, CR, PR, DDC, and DoR: up to 3 years.
Description: Reported safety data based upon the Intent-to-Treat Population: all enrolled participants who received at least 1 dose of SL-701.
Arm/Group | SL-701 + GM-CSF + Imiquimod | SL-701 + Poly-ICLC + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 38/46 | 16/28
Serious Adverse Events (participants affected / at risk) | 14/46 | 9/28
Other Adverse Events (participants affected / at risk) | 42/46 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SL-701 + GM-CSF + Imiquimod (N=46) | SL-701 + Poly-ICLC + Bevacizumab (N=28)
Vision blurred (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seizure (Nervous system disorders) | 4 | 2
Hemiparesis (Nervous system disorders) | 4 | 0
Encephalopathy (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 3 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 1
Mania (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | SL-701 + GM-CSF + Imiquimod (N=46) | SL-701 + Poly-ICLC + Bevacizumab (N=28)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 9 | 6
Vomiting (Gastrointestinal disorders) | 8 | 4
Constipation (Gastrointestinal disorders) | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 11 | 17
Injection site reaction (General disorders) | 7 | 8
Gait disturbance (General disorders) | 5 | 7
Injection site erythema (General disorders) | 7 | 4
Injection site pain (General disorders) | 2 | 7
Influenza like illness (General disorders) | 3 | 4
Injection site induration (General disorders) | 7 | 0
Chills (General disorders) | 4 | 1
Injection site swelling (General disorders) | 4 | 1
Injection site rash (General disorders) | 3 | 1
Asthenia (General disorders) | 1 | 2
Pyrexia (General disorders) | 3 | 0
Candida infection (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 1 | 2
Herpes zoster (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 5 | 9
Blood lactate dehydrogenase increased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Headache (Nervous system disorders) | 10 | 11
Aphasia (Nervous system disorders) | 7 | 6
Hemiparesis (Nervous system disorders) | 8 | 4
Seizure (Nervous system disorders) | 5 | 2
Dizziness (Nervous system disorders) | 3 | 3
Cognitive disorder (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 3 | 2
Memory impairment (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 2 | 2
Amnesia (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 3 | 0
Confusional state (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 5 | 2
Anxiety (Psychiatric disorders) | 3 | 3
Depression (Psychiatric disorders) | 1 | 3
Abulia (Psychiatric disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 2 | 6
Haematuria (Renal and urinary disorders) | 2 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Skin induration (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Hypertension (Vascular disorders) | 2 | 9
Sinus tachycardia (Cardiac disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 2 | 1
Blepharospasm (Eye disorders) | 1 | 0
Conjunctival irritation (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1
Mydriasis (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Injection site bruising (General disorders) | 0 | 1
Injection site discomfort (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Injection site cellulitis (Infections and infestations) | 1 | 0
Injection site infection (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Eye contusion (Injury, poisoning and procedural complications) | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Drug level decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Overweight (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 | 0
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 2 | 1
Ataxia (Nervous system disorders) | 1 | 1
Disturbance in attention (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 1
Facial paresis (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0
Apraxia (Nervous system disorders) | 0 | 1
Clumsiness (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Fine motor delay (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Muscular weakness (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Frustration tolerance decreased (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1
Hyposomnia (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 2 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0/30 | 1/18 — This adverse event affected only male participants.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Induration (General disorders) | 2 | 1
Injection site pruritus (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-10): https://cdn.clinicaltrials.gov/large-docs/48/NCT02078648/Prot_002.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT02078648/SAP_003.pdf